CLINICAL TRIAL: NCT03679962
Title: Adjunctive Triple Chronotherapy in the Acute Treatment of Depression and Suicidality in the Adolescent Population: A Randomized Controlled Trial
Brief Title: Triple Chronotherapy in Adolescents
Acronym: TCT-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Billings Clinic (Other)
Responsible Party: Principal Investigator, Mariela Herrera, Principal Investigator, Billings Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18.26
Record Dates: First submitted 2018-08-24; First posted 2018-09-21 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2022-07

CONDITIONS: Depressive Disorder, Major; Bipolar Depression; Suicidal Ideation
Keywords: Bright Light Therapy; Sleep Deprivation; Adolescent; Depression; Suicidal Ideation
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Suicidal Ideation; Sleep Deprivation; Depression | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triple Chronotherapy (Experimental): Four-day intervention, with 24-hour total sleep deprivation, 3-days of sleep phase advancement and daily bright light therapy.
  Interventions: Behavioral: Triple Chronotherapy
- Treatment as Usual (Active Comparator): Normal inpatient care, including pharmacotherapy, psychotherapy, milieu therapy and social work interventions
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Triple Chronotherapy — Day 0: One night of total sleep deprivation. The first 24 hours are spent with 1:1 nursing care for provision of comfort measures to stimulate wakefulness and to encourage completion of the intervention.
  Day 1-4: Sleep phase advancement Day 1: Sleep from 6 PM to 1 AM Day 2: Sleep from 8 PM to 3 AM Day 3: Sleep from 10 PM and 5 AM Day 4: Awaken at 5 AM; discharge following light therapy
  On days 1-4 patients will receive bright light therapy at 7am to 7:30am using a 10,000 Verilux light box. At discharge patients will be given a light box, strongly advised to continue the maintenance sleep schedule and bright light therapy at 7am daily for 30 minutes. Patients will be scheduled for follow-up appointments at 1-week, 1-month and 2-month following discharge.
  Arms: Triple Chronotherapy
Behavioral: Treatment as Usual — Normal inpatient care, including pharmacotherapy, psychotherapy, milieu therapy and social work interventions
  Arms: Treatment as Usual

SUMMARY:
Study Purpose This study is a randomized controlled trial examining the effectiveness of TCT in the acute treatment of depression and suicidality in adolescents compared to usual treatment care, which includes individual and group therapy, and medication adjustments. All potential participants will be identified at admission to the Psychiatric Youth Inpatient Unit of Billings Clinic and invited to participate. The length of participation is 2 months.

Study Design The primary research question of this RCT is whether adjunctive TCT in depressed adolescents is more effective in the management of depression symptoms and in reducing suicidal ideation at two months follow-up, than those adolescents who are receiving usual care. A total of three aims are proposed.

Hypothesis: Adjunctive TCT is more effective in the management of depression symptoms and in reducing suicidal ideation at two month follow-up than those adolescents who are receiving usual care.

The first aim is to track the trajectories of depression symptoms, suicidal ideation, and insomnia severity in participants receiving TCT and in those receiving treatment as usual over 4 days of initial treatment, thereby answering the question of whether adjunctive TCT can effectively reduce the severity of depression, insomnia and suicidal ideation.

The second aim is to examine whether TCT is more effective than usual care in sustaining treatment effects to the end of study period (2 months follow-up), therefore answering the question whether the effectiveness of the 4-day intervention of adjunctive TCT arm is sustainable up to the end of a two-month follow-up.

Hypothesis: TCT is more effective than usual care in sustaining treatment effects to the end of the study period than usual care.

The third aim is to assess the link to the clinical outcomes (change in depression symptoms, suicidal ideation, insomnia severity, and disease-associated quality of life) and patient satisfaction with the treatment.

Hypothesis: Clinical outcomes (depression symptoms, suicidal ideation, insomnia, and disease-related quality of life) and patient satisfaction are more effective than usual care alone.

DETAILED DESCRIPTION:
According to the Centers for Disease Control, almost 11% of youth will have met criteria for a depressive disorder by the time they are 18 years of age. Depression can significantly impact quality of life and is associated with increased risk of suicide, the second leading cause of death among individuals between ages 10 -24 years. While evidence-based treatments for the management of depression in adolescents exist, social stigma, perception that depression can be self-managed without treatment and side effects of antidepressants all pose treatment barriers. Moreover, the two most widely used evidence-based treatments, antidepressants and cognitive behavioral therapy, have medium to small effect sizes, and a significant need exists to develop more effective strategies to manage depression in adolescents. Adjunctive treatments for depression such as electroconvulsive therapy, transcranial magnetic stimulation, and ketamine have been shown to be effective in producing an antidepressant response in the adult population; however, none are yet recommended for safe use in adolescents. Moreover, ketamine and electroconvulsive therapy are associated with significant side effects, making each a less desirable treatment for depression among adolescent patients and their families.

Chronotherapy, defined as the therapeutic manipulation of sleep-wake cycles, is a promising approach for the treatment of adolescent depression. The study of chronotherapeutic interventions as an adjunctive treatment for depression began in the 1970s, when investigators noted a rapid, albeit transient, antidepressant response to sleep deprivation. Another chronotherapeutic technique, bright light therapy, has consistently shown benefit in the treatment of seasonal affective disorders. Its use in the treatment of non-seasonal unipolar and bipolar depression has also shown promising results.

Combination chronotherapeutics, such as triple chronotherapy (TCT), have also been trialed with some demonstrated efficacy. TCT is an approach that combines sleep deprivation, bright light therapy, and sleep phase advancement in the acute treatment of depression. One of the first open label TCT studies enrolled 143 consecutive patients; of the 141 adults who completed the study, a significant acute antidepressant response was found in up to 70% of patients with bipolar depression, and a sustained response in up to 55% of patients at 1-month. A more recent randomized control trial of 75 adults employed an abbreviated protocol that included one night of sleep deprivation, three nights of sleep phase advancement, and bright light therapy in each of the four mornings of the intervention. This study demonstrated similar, accelerated antidepressant responses along with a decrease in suicidality and improved sleep quality.

Although evidence is growing for the use of TCT to manage acute depression and suicidality in adults, studies in the adolescent population are lacking. It was hypothesized by Gest et al. (2014) that the use of chronotherapy in adolescents could be an effective treatment modality, and researchers were urged to explore this area. In 2016, Gest et al. compared combined sleep deprivation and bright light therapy to bright light therapy alone in adolescents and found a significant antidepressant response to bright light therapy alone, but no significant benefit was gained with the addition of one night of total sleep deprivation. Sleep phase advancement was absent in this study. No studies were found that examined the use of comprehensive TCT in adolescents compared to usual practice in the inpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be 12-17 years of age
* Must verbalize motivation for treatment
* Must provide informed assent; parent or guardian must provide consent
* Must be diagnosed with moderate to severe unipolar or bipolar depression. Severity of depression is determined using the Patient Health Questionnaire-9 (PHQ-9 modified for Adolescents [PHQ-A]). A score of 10 or more indicates moderate-severe depression

Exclusion Criteria:

* Active psychosis
* Manic state
* Younger than 12 years of age or older than 17 years of age
* Seizure disorder
* Pregnancy
* Lack of assent and consent
* Previous TCT treatment

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-03-14 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire -Adolescent version (PHQ-A) | PHQ-A the day prior to total sleep deprivation, and then again over the next 3 consecutive days.
  Measuring the change score of pre-post PHQ-A; a score of 5-9 indicates mild depression with watchful waiting and repeat test, 10-14 indicates moderate depression that should be followed up with due consideration as to counseling and/or pharmacotherapy, 15-19 signifies moderately severe depression what requires initiation of pharmacotherapy and/or psychotherapy, and a score of 20-27 is interpreted as severe depression with immediate initiation of pharmacotherapy and referral to a mental health specialist for psychotherapy and collaborative management.
Columbia Suicide Severity Rating Scale | Daily throughout the treatment (Days 0-4)
  Measuring the change score of pre-post C-SSRS; 5 potential questions- yes/no questions indicating suicidal behavior and ideation; optimum score = 0.

SECONDARY OUTCOMES:
Patient Health Questionnaire-Adolescent version (PHQ-A) | PHQ-A the day prior to total sleep deprivation, and then again over the next 3 consecutive days, at 1-month and at 2-month
  Measuring the change score of pre-post PHQ-A; a score of 5-9 indicates mild depression with watchful waiting and repeat test, 10-14 indicates moderate depression that should be followed up with due consideration as to counseling and/or pharmacotherapy, 15-19 signifies moderately severe depression what requires initiation of pharmacotherapy and/or psychotherapy, and a score of 20-27 is interpreted as severe depression with immediate initiation of pharmacotherapy and referral to a mental health specialist for psychotherapy and collaborative management
Youth Quality of life Questionnaire | Day 0 and repeat measure at 30 days
  Youth Quality of Life Instrument-Short Form (YQOL-SF); 16-questions each having a 0-10 score, higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Mariela Herrera, MD, Principal Investigator — Billings Clinic; Laurie Riemann, BSN, Study Director — Billings Clinic; Jamie Besel, MSN, Study Chair — Billings Clinic
Locations (1):
- Billings Clinic, Billings, Montana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heron M. Deaths: Leading Causes for 2014. Natl Vital Stat Rep. 2016 Jun;65(5):1-96. PMID 27376998
- [Background] Gulliver A, Griffiths KM, Christensen H. Perceived barriers and facilitators to mental health help-seeking in young people: a systematic review. BMC Psychiatry. 2010 Dec 30;10:113. doi: 10.1186/1471-244X-10-113. PMID 21192795
- [Background] Abdallah CG, Adams TG, Kelmendi B, Esterlis I, Sanacora G, Krystal JH. KETAMINE'S MECHANISM OF ACTION: A PATH TO RAPID-ACTING ANTIDEPRESSANTS. Depress Anxiety. 2016 Aug;33(8):689-97. doi: 10.1002/da.22501. Epub 2016 Apr 6. PMID 27062302
- [Background] Cao B, Luo Q, Fu Y, Du L, Qiu T, Yang X, Chen X, Chen Q, Soares JC, Cho RY, Zhang XY, Qiu H. Predicting individual responses to the electroconvulsive therapy with hippocampal subfield volumes in major depression disorder. Sci Rep. 2018 Apr 3;8(1):5434. doi: 10.1038/s41598-018-23685-9. PMID 29615675
- [Background] Kayser S, Bewernick BH, Wagner S, Schlaepfer TE. Clinical Predictors of Response to Magnetic Seizure Therapy in Depression: A Preliminary Report. J ECT. 2019 Mar;35(1):48-52. doi: 10.1097/YCT.0000000000000495. PMID 29613946
- [Background] Pflug B, Tolle R. Disturbance of the 24-hour rhythm in endogenous depression and the treatment of endogenous depression by sleep deprivation. Int Pharmacopsychiatry. 1971;6(3):187-96. doi: 10.1159/000468269. No abstract available. PMID 4950570
- [Background] Nussbaumer B, Kaminski-Hartenthaler A, Forneris CA, Morgan LC, Sonis JH, Gaynes BN, Greenblatt A, Wipplinger J, Lux LJ, Winkler D, Van Noord MG, Hofmann J, Gartlehner G. Light therapy for preventing seasonal affective disorder. Cochrane Database Syst Rev. 2015 Nov 8;(11):CD011269. doi: 10.1002/14651858.CD011269.pub2. PMID 26558494
- [Background] Tuunainen A, Kripke DF, Endo T. Light therapy for non-seasonal depression. Cochrane Database Syst Rev. 2004;2004(2):CD004050. doi: 10.1002/14651858.CD004050.pub2. PMID 15106233
- [Background] Al-Karawi D, Jubair L. Bright light therapy for nonseasonal depression: Meta-analysis of clinical trials. J Affect Disord. 2016 Jul 1;198:64-71. doi: 10.1016/j.jad.2016.03.016. Epub 2016 Mar 15. PMID 27011361
- [Background] Benedetti F, Riccaboni R, Locatelli C, Poletti S, Dallaspezia S, Colombo C. Rapid treatment response of suicidal symptoms to lithium, sleep deprivation, and light therapy (chronotherapeutics) in drug-resistant bipolar depression. J Clin Psychiatry. 2014 Feb;75(2):133-40. doi: 10.4088/JCP.13m08455. PMID 24345382
- [Background] Martiny K, Refsgaard E, Lund V, Lunde M, Sorensen L, Thougaard B, Lindberg L, Bech P. A 9-week randomized trial comparing a chronotherapeutic intervention (wake and light therapy) to exercise in major depressive disorder patients treated with duloxetine. J Clin Psychiatry. 2012 Sep;73(9):1234-42. doi: 10.4088/JCP.11m07625. PMID 23059149
- [Background] Martiny K, Refsgaard E, Lund V, Lunde M, Thougaard B, Lindberg L, Bech P. Maintained superiority of chronotherapeutics vs. exercise in a 20-week randomized follow-up trial in major depression. Acta Psychiatr Scand. 2015 Jun;131(6):446-57. doi: 10.1111/acps.12402. Epub 2015 Feb 17. PMID 25689725
- [Background] Gest S, Legenbauer T, Bogen S, Schulz C, Pniewski B, Holtmann M. Chronotherapeutics: an alternative treatment of juvenile depression. Med Hypotheses. 2014 Mar;82(3):346-9. doi: 10.1016/j.mehy.2014.01.002. Epub 2014 Jan 15. PMID 24468576
- [Background] Gest S, Holtmann M, Bogen S, Schulz C, Pniewski B, Legenbauer T. Chronotherapeutic treatments for depression in youth. Eur Child Adolesc Psychiatry. 2016 Feb;25(2):151-61. doi: 10.1007/s00787-015-0720-6. Epub 2015 May 17. PMID 25982568
- See also: National Institute of Mental Health. Mental Health Information. 2015 — http://www.nimh.nih.gov/health/topics/index.shtml